CLINICAL TRIAL: NCT02998151
Title: Neurophysiological and Acute Pharmacological Studies in FXS Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CIN001 - {LAM}; U54HD082008 (NIH)
Record Dates: First submitted 2016-12-01; First posted 2016-12-20 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Acamprosate; Lovastatin; Minocycline; Baclofen

STUDY DESIGN:
Intervention Model Description: This study was designed as a 4-intervention crossover, with all study participants receiving all possible interventions. These were originally placebo, acamprosate, minocycline, and lovastatin. Midway through the study (n=16) it was determined that acamprosate was undetectable in serum and this intervention was replaced by baclofen. Remaining participants (n=13) received baclofen and 5 participants were re-enrolled to receive baclofen or a second round of placebo, so investigators and participants would remain blinded to drug status during the baclofen visit. The second round of placebo was not analyzed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- All Study Participants (Experimental): Participants received, in random order, a single dose of placebo, acamprosate, lovastatin, minocycline, or baclofen, with a two-week washout period between doses. Midway through the study (n=16) it was determined that acamprosate was undetectable in serum and this intervention was replaced by baclofen. Remaining participants (n=13) received baclofen and 5 participants were re-enrolled to receive baclofen or a second round of placebo, so investigators and participants would remain blinded to drug status during the baclofen visit. The second round of placebo was not analyzed.
  Interventions: Drug: Acamprosate; Drug: Lovastatin; Drug: Minocycline; Drug: Placebo; Drug: Baclofen

INTERVENTIONS:
Drug: Acamprosate — two 666mg pills
Drug: Lovastatin — two 20mg pills
Drug: Minocycline — two 135mg pills
Drug: Placebo — placebo pill
Drug: Baclofen — one 30mg pill

SUMMARY:
The aim of this study is to utilize neurophysiologic assessments, behavioral measures and clinical measures to assess how much deficits associated with Fragile X Syndrome from pre-dose to post-dose using pharmacology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 15-55, with fragile X syndrome (FXS) who completed the study entitled "Mechanisms and brain circuits underlying fragile X syndrome (IRB # 2015-8425). FXS is defined as full FMR1 mutations (>200 CGG repeats) confirmed by genetic testing.
* General good health as determined by physical exam, medical history and laboratory work up.

Exclusion Criteria:

* Subjects with a history of intolerance to acamprosate, lovastatin, or minocycline will be excluded.
* Subjects will also be excluded if they have taken any investigational drug within 3 months, have a history of substance abuse or dependence within 6 months, or significant psychiatric or central nervous system neurological disease unrelated to FXS.
* Uncontrolled seizures impact EEG data as do anticonvulsants, barbiturates, lithium and benzodiazepines and are exclusions (within 5 half-lives). Those taking other psychiatric medications must be on stable doses for 4 weeks before any testing.
* For female subjects of child bearing potential, a positive urine pregnancy test.
* Potential subjects with a creatinine clearance < 50 mL/min will be excluded.
* Identified medical issues, inability to tolerate study procedures or study drug per the discretion of the Principal Investigator.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Erickson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Jonak CR, Pedapati EV, Schmitt LM, Assad SA, Sandhu MS, DeStefano L, Ethridge L, Razak KA, Sweeney JA, Binder DK, Erickson CA. Baclofen-associated neurophysiologic target engagement across species in fragile X syndrome. J Neurodev Disord. 2022 Sep 27;14(1):52. doi: 10.1186/s11689-022-09455-9. PMID 36167501

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants engaged in a baseline visit to gather preliminary data and ensure study compliance. Participants were then randomly assigned to different sequences for receiving acamprosate, lovastatin, minocycline, baclofen, and placebo. There was a 2-week washout period between visits.
Groups:
- All Study Participants: This study was designed as a 4-intervention crossover, with all study participants receiving all possible interventions. These were originally placebo, acamprosate, minocycline, and lovastatin. Midway through the study (n=16) it was determined that acamprosate was undetectable in serum and this arm was replaced by baclofen. Remaining participants (n=13) received baclofen and 5 participants were re-enrolled to receive baclofen.
Period: Overall Study
Arm/Group | All Study Participants
Started | 29
Placebo | 27 (Two participants withdrew from the study before receiving placebo.)
Acamprosate (Acamprosate was discontinued due to undetectable serum levels after dosage.) | 16 (Every participant received acamprosate prior to acamprosate's discontinuance.)
Lovastatin | 29 (All participants received lovastatin.)
Minocycline | 27 (Two participants withdrew from the study before receiving minocycline.)
Baclofen (Baclofen replaced acamprosate after it was determined acamprosate was undetectable in serum after dosage.) | 18 (All 13 remaining participants received baclofen after acamprosate was discontinued. Five participants were re-enrolled to receive baclofen.)
Completed (Five participants completed all 5 study arms; however, 26 completed all that were originally asked of them (4 visits, with 5 of those 26 re-enrolling to complete baclofen as well).) | 5 (Acamprosate was discontinued mid-study due to undetectable serum levels and replaced with baclofen. Participants who already completed acamprosate were given the option to re-enroll and receive baclofen. Five participants received all 5 interventions; 26 received 4+ interventions.)
Not Completed | 24
Not completed — Withdrawal by Subject | 3
Not completed — Participant declined to re-enroll for baclofen | 8
Not completed — Participant was not offered acamprosate; acamprosate was discontinued and replaced with baclofen | 13

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.71 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 29
Woodcock Johnson Test of Cognitive Abilities - Auditory Attention Task [Mean (Standard Deviation); unit: scores on a scale] — Measure Description: Woodcock Johnson Test of Cognitive Abilities III Auditory Attention subscale. Participants must identify orally presented words amid increasingly intense background noise. The scores for this subtask range from 0-50, with higher scores indicating a better outcome. Raw scores for this subscale are reported (rather than standard scores, or age- or grade-equivalents). Population: One participant did not complete the Woodcock Johnson.
  scores on a scale
    number analyzed (Participants) | 28
    (all) | 30.89 (4.92)

OUTCOME MEASURES:

1. Primary Outcome: Change in EEG Relative Gamma Power
Description: EEG relative gamma power at rest was calculated as the percent of power in the gamma frequencies relative to the sum of power in all frequency bands, averaged across electrodes, and calculated separately at pre-dose and post-dose timepoints. To assess the impact of drug, the pre-dose relative gamma power was subtracted from post-dose relative gamma power. Higher numbers indicate more relative gamma power post-dose; lower numbers indicate more relative gamma power pre-dose.
Time Frame: Pre-dose, 4-hour post-dose
Population: Missing 1 placebo, 1 lovastatin who contributed data with excessive movement or other artifact, or were unable to complete the task.
Measure: Mean (Standard Deviation); unit: percent of power in gamma frequencies
Arm/Group | Placebo | Acamprosate | Lovastatin | Minocycline | Baclofen
Number analyzed (Participants) | 26 | 16 | 28 | 27 | 18
percent of power in gamma frequencies | 0.0024 (.0265) | -0.0077 (0.0252) | -0.0039 (0.0225) | 0.0019 (0.0235) | -0.0160 (0.0346)

2. Primary Outcome: Clinical Global Impressions-Improvement
Description: The Clinical Global Impressions - Improvement (CGI-I) requires the clinician to assess how much the patient's illness has changed relative to pre-dose, from 1 (very much improved) to 7 (very much worse).
Time Frame: 4-hour post-dose
Population: CGI-I was not collected for one participant on their minocycline day and another participant on their baclofen day.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acamprosate | Lovastatin | Minocycline | Baclofen
Number analyzed (Participants) | 27 | 16 | 29 | 26 | 17
score on a scale | 3.70 (.61) | 3.88 (.62) | 3.97 (.50) | 3.81 (.49) | 3.94 (.43)

3. Secondary Outcome: Woodcock Johnson Test of Cognitive Abilities - Auditory Attention Task
Description: Woodcock Johnson Test of Cognitive Abilities III Auditory Attention subscale. Participants must identify orally presented words amid increasingly intense background noise. The scores for this subtask range from 0-50, with higher scores indicating a better outcome. Raw scores for this subscale are reported (rather than standard scores, or age- or grade-equivalents).
Time Frame: 4-hour post-dose
Population: Data is missing from 2 placebo, 1 acamprosate, 1 lovastatin, 2 minocycline, and 1 baclofen.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acamprosate | Lovastatin | Minocycline | Baclofen
Number analyzed (Participants) | 25 | 15 | 28 | 25 | 17
score on a scale | 32.84 (5.77) | 33.07 (5.48) | 32.93 (5.31) | 33.24 (6.04) | 33 (5.17)

4. Secondary Outcome: Change From Pre-dose in the Repeatable Battery for the Assessment of Neuropsychological Status at 4 Hours Post Dose
Description: Four 10-item lists of unrelated words were presented orally to the examinee who was then required to immediately recall words presented, at both pre-dose and post-dose timepoints. The impact of drug was assessed by subtracting the number of words remembered post-dose from the number of words remembered pre-dose. Lower numbers indicate more words remembered post-dose; higher numbers indicate more words remembered pre-dose.
Time Frame: Pre-dose, 4-hour post dose
Population: One participant is missing from placebo, acamprosate, lovastatin, and minocycline conditions due to being unable to repeat list words back to experimenter (nonverbal). Baclofen and placebo are each additionally missing one participant who did not complete the pre-dose or post-dose task.
Measure: Mean (Standard Deviation); unit: number of words remembered
Arm/Group | Placebo | Acamprosate | Lovastatin | Minocycline | Baclofen
Number analyzed (Participants) | 25 | 15 | 28 | 26 | 17
number of words remembered | -.20 (4.23) | -1.47 (5.17) | -1.25 (3.85) | -.69 (5.58) | -.88 (3.35)

5. Secondary Outcome: Test of Attentional Performance for Children (KiTAP) Test of Alertness
Description: Computerized task where an examinee is required to push a key when a target stimulus is presented on the screen. Scores are presented as change in median reaction time (RT), in milliseconds.
Time Frame: Predose, 4-hour post-dose
Population: One participant is missing from the placebo, acamprosate, lovastatin, and minocycline conditions due to being unable to participate in the task. An additional one participant each is missing from placebo, acamprosate, and lovastatin conditions due to uncollected data at either the pre-dose or post-dose timepoint.
Measure: Mean (Standard Deviation); unit: change in median RT in milliseconds
Arm/Group | Placebo | Acamprosate | Lovastatin | Minocycline | Baclofen
Number analyzed (Participants) | 25 | 14 | 27 | 26 | 18
change in median RT in milliseconds | 13.76 (188.37) | -28.64 (137.21) | 18.59 (169.39) | 26.85 (226.69) | -31.44 (171.91)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to four weeks after the final dosing visit.
Description: Participants were asked about adverse events in person 4 hours after each dose and at the end of each dosing visit, and via phone calls conducted one day after and 8 days after each dosing visit. Additionally, participants were contacted by phone 4 weeks after the final dosing visit.
Arm/Group | Placebo | Acamprosate | Lovastatin | Minocycline | Baclofen
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/16 | 0/29 | 0/27 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/16 | 0/29 | 0/27 | 0/18
Other Adverse Events (participants affected / at risk) | 3/27 | 7/16 | 4/29 | 4/27 | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Acamprosate (N=16) | Lovastatin (N=29) | Minocycline (N=27) | Baclofen (N=18)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — excessive talking or hyperactivity
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Latest study protocol with baclofen (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT02998151/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Previous study protocol with original arms (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02998151/Prot_SAP_001.pdf
  • Informed Consent Form: Latest consent form with baclofen (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02998151/ICF_002.pdf